CLINICAL TRIAL: NCT02880670
Title: Pharmacokinetics and Metabolism of [14C] BMS-986142 in Healthy Male Subjects
Brief Title: Pharmacokinetics and Metabolism Study of Radiolabeled BMS-986142 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM006-022
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Arthritis
Keywords: Rheumatoid
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose of radiolabeled BMS-986142 (Experimental)
  Interventions: Drug: BMS-986142

INTERVENTIONS:
Drug: BMS-986142

SUMMARY:
This is an open-label, single-dose, study in healthy males. The primary objective is to assess the pharmacokinetics (PK), metabolism, and routes of elimination of a single oral dose of radiolabeled BMS-986142 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Target population: Healthy males with no clinically significant deviations from normal in medical history, physical examinations, vital signs, electrocardiograms (ECGs), physical measurements, and clinical laboratory tests
* Body weight of at least 50 kilograms (110 pounds); body mass index (BMI) between 18 to 32 kg/m2.

Exclusion Criteria:

* History of any chronic or acute illness including active TB in the last 3 years, recent infection, gastrointestinal disease, smoking within less than 6 months prior to dosing, alcohol abuse, inability to tolerate oral medication, or inability to be venipunctured.
* Vaccination or plans for vaccination with any live vaccine 12 weeks prior to first dose of study drug, during the course of the study, or 30 days after the last dose of study drug.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiograms, or clinical laboratory determinations beyond what is consistent with the target population.
* History of allergies and adverse drug reaction to any oral contraceptive compounds or Bruton tyrosine kinase (BTK) inhibitors.
* Participated in a radiolabeled drug study within the previous 12 months; clinically significant diagnostic or therapeutic radiation exposure within the previous 12 months; or current employment in a job requiring radiation exposure monitoring.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is PK parameters that will be determined from plasma concentration versus time | Day 1 to Day 13
Urinary/fecal/bile (if applicable) TRA (Total radioactivity) recovery data | Day 1 to Day 13

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and the results of electrocardiogram tests (ECGs), vital signs, physical exams, and clinical laboratory tests. | Day 1 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx